CLINICAL TRIAL: NCT05429658
Title: A Prospective, Single-arm, Interventional Clinical Trial to Evaluate the Safety and Effectiveness of the Route 92 Medical MonoPoint Reperfusion System for Aspiration Embolectomy in Acute Ischemic Stroke Patients
Brief Title: Single Arm Trial to Evaluate the Safety and Effectiveness of the Route 92 Medical Reperfusion System
Acronym: SUMMITNZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Route 92 Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CIP 0605
Record Dates: First submitted 2022-06-16; First posted 2022-06-23 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2022-06

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Thrombectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Thrombectomy (Experimental): Aspiration of clot with large bore catheter in acute ischemic stroke patients
  Interventions: Device: Thrombectomy

INTERVENTIONS:
Device: Thrombectomy — The Route 92 Medical Reperfusion System is indicated for use in the revascularization of patients with acute ischemic stroke secondary to intracranial large vessel occlusive disease within the internal carotid, middle cerebral, basilar and vertebral arteries.

SUMMARY:
The objective of the study is to evaluate the safety and effectiveness of the Route 92 Medical Monopoint Reperfusion System with the Hi Point 88 and HiPoint 70 Reperfusion Catheters when used to aspirate emboli in acute ischemic stroke patients.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the safety and effectiveness of the Route 92 Medical Monopoint Reperfusion System with the Hi Point 88 and HiPoint 70 Reperfusion Catheters when used to aspirate emboli in acute ischemic stroke patients.

The study design is an interventional, prospective, single-arm, open label clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. The consent process has been completed with the subject, Legally Authorized Representative, or two physician best interest and consent is documented
2. Age >18 years
3. Clinical signs consistent with an acute ischemic stroke
4. Baseline National Institutes of Health Stroke Scale (NIHSS) score >= 6
5. Pre-stroke modified Rankin Score (mRS) <= 2
6. Acute occlusion of the M1 segment of the middle cerebral artery (MCA), internal carotid artery (ICA), vertebral or basilar arteries confirmed via computed tomography angiography (CTA) and/or magnetic resonance angiography (MRA)
7. The Investigator estimates that at least one delivery of the Route 92 Medical Reperfusion System can be completed within 24 hours of time last known well
8. In the opinion of the Investigator, reperfusion of the ischemic territory will result in clinical benefit
9. Angiographic confirmation of an occlusion of the M1 segment* of the middle cerebral artery, internal carotid artery, vertebral or basilar arteries with a modified Thrombolysis In Cerebral Infarction (mTICI) scale score of 0-1

Exclusion Criteria:

1. Known pregnancy or breast feeding
2. Known comorbidity that may complicate treatment or prevent improvement or follow-up
3. Known life expectancy < 12 months
4. Known history of severe allergy to contrast medium
5. Subject known to have suffered a stroke in the past 90 days
6. Subject participating in another study involving an investigational device or drug.
7. Known connective tissue disorder affecting the arteries (e.g. Marfan syndrome, fibromuscular dysplasia, Ehlers-Danlos syndrome)
8. Any known pre-existing hemorrhagic or coagulation deficiency
9. Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) evidence of recent/ fresh hemorrhage
10. Baseline CT or MRI showing intracranial tumor (except small meningioma)
11. Angiographic evidence of dissection in the extracranial or intracranial arteries
12. Angiographic evidence of carotid dissection
13. Angiographic evidence of multiple vascular occlusions (e.g., bilateral anterior circulation, anterior/posterior circulation). Note: tandem occlusions may be included at the discretion of the operating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Effectiveness | Procedure
  The primary effectiveness endpoint is arterial revascularization as measured by a modified Thrombolysis in Cerebrovascular Infarction (mTICI) score of 2b or greater at the end of angiography after all endovascular treatments.
Device-related peri-procedural complications | Procedure
  dissection or perforation
Symptomatic Intracranial Cerebral Hemorrhage (SICH) | 24 hour
  defined as type 2 parenchymal hemorrhage with a deterioration in National Institutes of Health Stroke Scale [NIHSS] score of >=4 points
Embolization to a previously uninvolved territory | Procedure
  Embolization to a previously uninvolved territory

SECONDARY OUTCOMES:
NIHSS score | 24 hours after treatment
  The National Institutes of Health Stroke Scale (NIHSS) is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke
Modified Rankin Score | 90 days after treatment
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or who have other causes of neurological disability
Procedure Time | Procedure
  Total procedure time from insertion of Route 92 Reperfusion System to final angiogram
Procedure-Related SAEs | Procedure
  Serious Adverse Events related to the interventional procedure

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Brew, MBChB, MHB, Principal Investigator — Auckland City Hospital
Locations (2):
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch

IPD SHARING:
Plan to Share IPD: No